CLINICAL TRIAL: NCT04060940
Title: Emotion Regulation Therapy for Young Adults With Clinical Worry and Rumination
Brief Title: Emotion Regulation Therapy for Clinical Worry and Rumination
Acronym: ERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Douglas Mennin (Other)
Collaborators: Kent State University (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor-Investigator, Douglas Mennin, Professor of Clinical Psychology, Teachers College, Columbia University
Organization: Teachers College, Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-019
Record Dates: First submitted 2019-06-04; First posted 2019-08-19 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Anxiety Disorders and Symptoms; Depression, Anxiety; Generalized Anxiety Disorder; Emotional Dysfunction
Keywords: Emotion Regulation; Distress Disorders; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression; Generalized Anxiety Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: All participants will be randomly assigned to an 8-session or 16-session version of ERT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Regulation Therapy: 8-session version (Experimental): All participants will be randomly assigned to an 8-session or 16-session version of ERT with equal probability. Participants assigned to the 8-session version of ERT will receive 8 sessions of individualized therapy, each of which is 1-1.5 hours, on a weekly basis. Sessions 1-5 will be 1 hour long, sessions 6 and 7 will be 1.5 hours long, and session 8 will be one hour long, resulting in a total required time commitment of 9 hours over the course of 8 weeks.
  Interventions: Behavioral: Emotion Regulation Therapy: 8-session version
- Emotion Regulation Therapy: 16-session version (Experimental): All participants will be randomly assigned to an 8-session or 16-session version of ERT with equal probability. Participants assigned to the 16-session version of ERT will receive 16 sessions of individualized therapy, each of which is 1-1.5 hours, on a weekly basis. Sessions 1-9 will be 1 hour long, sessions 10-13 will be 1.5 hours long, and sessions 14-16 will be 1 hour long, resulting in a total required time commitment of 18 hours over the course of 16 weeks.
  Interventions: Behavioral: Emotion Regulation Therapy: 16-session version

INTERVENTIONS:
Behavioral: Emotion Regulation Therapy: 8-session version — Emotion Regulation Therapy will be administered over 8 individual sessions on a weekly basis, resulting in a total required time commitment of 9 hours over the course of 8 weeks. The initial stage of treatment focuses on psychoeducation about anxiety and depression, individual patterns of these behaviors, emotions in recent situations, and self-monitoring of worry, anxiety, and depression. The sessions focus on the development of skills that help regulate one's emotional experience (i.e., recognizing emotions when they are happening, identifying the meaning of a given emotion experience, and soothing oneself in the context of negative emotional experiences). Following the development of these skills, sessions focus on the application of somatic awareness and emotion regulation skills while imagining emotionally evocative themes. The remaining sessions focus on terminating therapy, relapse prevention, and future goals.
  Other Names: Emotion Regulation Therapy (ERT)
  Arms: Emotion Regulation Therapy: 8-session version
Behavioral: Emotion Regulation Therapy: 16-session version — Emotion Regulation Therapy will be administered over 16 individual sessions on a weekly basis, resulting in a total required time commitment of 18 hours over the course of 16 weeks. The initial stage of treatment focuses on psychoeducation about anxiety and depression, individual patterns of these behaviors, emotions in recent situations, and self-monitoring of worry, anxiety, and depression. The sessions focus on the development of skills that help regulate one's emotional experience (i.e., recognizing emotions when they are happening, identifying the meaning of a given emotion experience, and soothing oneself in the context of negative emotional experiences). Following the development of these skills, sessions focus on the application of somatic awareness and emotion regulation skills while imagining emotionally evocative themes. The remaining sessions focus on terminating therapy, relapse prevention, and future goals.
  Other Names: Emotion Regulation Therapy (ERT)
  Arms: Emotion Regulation Therapy: 16-session version

SUMMARY:
The present project aims to broaden our understanding of neural mechanisms which may underlie change in symptoms occurring over the course of Emotion Regulation Therapy. Specifically, we aim to examine neural changes as a result of either an 8-session or 16-session version of the treatment.

DETAILED DESCRIPTION:
This study aims to examine the utility of Emotion Regulation Training (ERT) in reducing symptoms of anxiety and/or depression in young adults aged 18 to 29 years old. Additionally, we are interested in assessing neural, cardiac, and immunological changes associated with psychological symptom reduction in these individuals. Lastly, we are interested in examining whether an abbreviated 8-session version of ERT produces similar results to a longer (16-session) version of ERT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-29 years during the time of participation
* Meets diagnostic criteria for an anxiety and/or depressive disorder
* Endorses significant worry and/or rumination

Exclusion Criteria:

* Active suicidal intent
* Current substance dependence disorder (within the past year)
* Current or past psychotic disorder, bipolar-I disorder, or dementia
* Not currently received any other form of psychosocial treatment
* Not being on a stabilized dose of medication (less than 3 months) during enrollment
* Pregnancy or plans to become pregnant during active participation
* Irremovable metal objects in the body
* Neurological disorder, traumatic brain injury, or loss of consciousness
* Tattoos if/when posing risks for involvement in the MRI component of the study

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Changes in Worry | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), Weekly for 8- or 16-weeks (depending on version), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Penn State Worry Questionnaire (PSWQ)
Changes in Rumination | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), Weekly for 8- or 16-weeks (depending on version), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Rumination-Reflection Questionnaire (RRQ)
Changes in Functional Impairment | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), Weekly for 8- or 16-weeks (depending on version), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Sheehan Disability Scale (SDS)
Changes in Life Satisfaction | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Quality of Life Inventory (QOLI)
Changes in Diagnostic Criteria, Severity, and Improvement | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Structured Clinical Interview for DSM-IV-TR; Clinical Severity Ratings from Anxiety Disorders Interview Schedule, Lifetime version for DSM-IV

SECONDARY OUTCOMES:
Changes in Anxiety and Depression | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Mood and Anxiety Symptom Questionnaire (MASQ)
Model-Related Changes: Attention Regulation | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), Weekly for 8- or 16-weeks (depending on version), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Attentional Control Scale (ACS)
Model-Related Changes: Metacognitive Regulation | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), Weekly for 8- or 16-weeks (depending on version), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Experiences Questionnaire (EQ); Emotion Regulation Questionnaire-Reappraisal (ERQ)

OTHER OUTCOMES:
Neural Changes using fMRI | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment)
  Resting State and Behavioral Tasks (i.e., Attentional Shifting Task, Emotion Regulation Task, Approach-Avoidance Conflict Task)
Cardiac Changes using HRV | Pre-Treatment, Mid-Treatment (either 4- or 8- weeks after starting treatment), Post-Treatment (either 8- or 16- weeks after starting treatment), 3-Month Follow-Up, 9-Month Follow-Up, 2-Year Follow-Up
  Resting State
Inflammatory Markers | Pre-Treatment, Post-Treatment (either 8- or 16- weeks after starting treatment)
  Blood Draw (i.e., IL-6, TNF-alpha, and the C-reactive protein)

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mennin DS, Fresco DM, O'Toole MS, Heimberg RG. A randomized controlled trial of emotion regulation therapy for generalized anxiety disorder with and without co-occurring depression. J Consult Clin Psychol. 2018 Mar;86(3):268-281. doi: 10.1037/ccp0000289. PMID 29504794
- [Result] Renna ME, Quintero JM, Soffer A, Pino M, Ader L, Fresco DM, Mennin DS. A Pilot Study of Emotion Regulation Therapy for Generalized Anxiety and Depression: Findings From a Diverse Sample of Young Adults. Behav Ther. 2018 May;49(3):403-418. doi: 10.1016/j.beth.2017.09.001. Epub 2017 Sep 8. PMID 29704969
- [Result] Renna ME, Quintero JM, Fresco DM, Mennin DS. Emotion Regulation Therapy: A Mechanism-Targeted Treatment for Disorders of Distress. Front Psychol. 2017 Feb 6;8:98. doi: 10.3389/fpsyg.2017.00098. eCollection 2017. PMID 28220089
- [Derived] Renna ME, Spaeth PE, Quintero JM, O'Toole MS, Sandman CF, Fresco DM, Mennin DS. A randomized controlled trial comparing two doses of emotion regulation therapy: Preliminary evidence that gains in attentional and metacognitive regulation reduce worry, rumination, and distress. Behav Res Ther. 2023 Oct 21;170:104420. doi: 10.1016/j.brat.2023.104420. Online ahead of print. PMID 39491310